CLINICAL TRIAL: NCT00724373
Title: Retrospective Data Study of HCV Genotype 1 Patients in the UK Treated With ViraferonPeg and Rebetol
Brief Title: Study of HCV Genotype 1 Patients in the UK Treated With ViraferonPeg and Rebetol (Study P05269)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05269
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2010-06-07 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with genotype 1 Hepatitis C Virus infection.: Participants with genotype 1 Hepatitis C Virus (HCV) infection who have been treated with pegylated interferon alfa-2b and ribavirin in the preceding 48 months
  Interventions: Biological: Peginterferon alfa-2b (SCH 54031); Drug: Ribavirin (SCH 18908)

INTERVENTIONS:
Biological: Peginterferon alfa-2b (SCH 54031) — Peginterferon alfa-2b plus ribavirin will be administered according to the products' labeling.
  Other Names: PegIntron; ViraferonPeg
Drug: Ribavirin (SCH 18908) — Peginterferon alfa-2b plus ribavirin will be administered according to the products' labeling.
  Other Names: Rebetol

SUMMARY:
The study is designed as a retrospective data review of medical records from participants selected from specialist secondary and tertiary care centers across the United Kingdom (UK), specializing in Hepatitis C treatment. The study is non-interventional and is designed to identify subgroups of Hepatitis C Virus (HCV) genotype 1 participants in the 'real world', including the relation between subgroup characteristics and treatment responsiveness.

DETAILED DESCRIPTION:
Physicians will record information (from the time of first exposure to pegylated interferon alfa-2b and ribavirin) from the medical notes of participants who fit the inclusion criteria. To prevent selection bias, data are to be taken from the latest consecutive, unique participants seen by the physician over the previous 48 months. This provides a method of random sampling from a physician practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with genotype 1 HCV infection who have been treated with pegylated interferon alfa-2b and ribavirin in the preceding 48 months will be included. They will be divided into:
* Completer participants: Patients with a diagnosis of HCV genotype 1 who have completed a course of interferon alfa-2b and ribavirin, with no prior treatment for HCV (ie, previously treatment naïve). Completer participants must have at least 24 weeks of follow up data available post completion of treatment to ensure ability to assess SVR rates.
* Early terminators: Participants who have terminated treatment early due to adverse events or other reasons (ie, exposure is incomplete).

Exclusion Criteria:

* Participants currently undergoing therapy and therefore have not terminated treatment, ie, exposure is still ongoing.
* Co-infected HCV participants (eg, human immunodeficiency virus [HIV] or hepatitis B virus [HBV]).
* Participants who received their first HCV treatment in relation to a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with genotype 1 HCV infection who have been treated with pegylated interferon alfa-2b and ribavirin in the preceding 48 months at sites in the UK.
Sampling Method: Probability Sample
Enrollment: 442 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Genotype 1 Hepatitis C Virus Infection.
Started | 442
Completed | 271
Not Completed | 171
Not completed — Adverse Event | 41
Not completed — Lack of Efficacy | 82
Not completed — Lost to Follow-up | 7
Not completed — Non-compliance | 2
Not completed — HCV RNA negative after 4 weeks | 9
Not completed — Participant moved away | 1
Not completed — Responder at 12 weeks, PCR + at 24 weeks | 2
Not completed — Only to have 24 week regimen | 1
Not completed — Viral Relapse | 1
Not completed — Acute HCV infection | 1
Not completed — Drug Relapse | 1
Not completed — Tolerability | 23

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Genotype 1 Hepatitis C Virus Infection.
Number analyzed (Participants) | 442
Age, Customized [Mean (Standard Deviation); unit: Years] — Mean age was calculated for 441 of the 442 participants. Age was missing for one participant.
  Years | 43 (10.13)
Sex/Gender, Customized [Number; unit: participants]
  Female | 143
  Male | 296
  Gender information missing | 3
Region of Enrollment [Number; unit: participants]
  United Kingdom | 442

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment Success
Description: Identify subgroups of genotype 1 participants to better understand factors affecting response rates & treatment outcomes & to provide predictive models of refractory or responsive phenotypes to aid in HCV treatment, management, & drug development. Treatment success is defined as those who had achieved sustained virological response (i.e. undetectable viraemia 24 weeks post therapy completion).
Time Frame: Data will be collected from the start of first exposure to pegylated interferon alfa-2b and ribavirin combination therapy. Participants who have successfully completed treatment will have data collected for a follow-up period of at least 24 weeks.
Population: Number of participants who had treatment success.
Measure: Number; unit: Participants
Arm/Group | Participants With Genotype 1 Hepatitis C Virus Infection.
Number analyzed (Participants) | 243
Participants
  Genotype 1a | 117
  Genotype 1b | 63
  Genotype 1a and 1b | 4
  Genotype 1c | 0
  Genotype 1 subgroup unspecified | 59

ADVERSE EVENTS:
Arm/Group | Pegylated Interferon Alfa-2b and Ribavirin
Serious Adverse Events (participants affected / at risk) | 17/442
Other Adverse Events (participants affected / at risk) | 0/442
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon Alfa-2b and Ribavirin (N=442)
ANAEMIA (Blood and lymphatic system disorders) | 4 (5)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2)
ANGINA PECTORIS (Cardiac disorders) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (2)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
SARCOIDOSIS (Immune system disorders) | 1 (1)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
ACUTE PSYCHOSIS (Psychiatric disorders) | 4 (4)
ANXIETY (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
HALLUCINATION (Psychiatric disorders) | 1 (1)
PARANOIA (Psychiatric disorders) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data will be the property of the Sponsor. Although under no obligation, it is asked that the investigator discuss any publication with the sponsor prior to release and obtain written consent. The sponsor recognises the right of the investigator to publish the results upon study completion. However, it is asked that the investigator send a draft to the sponsor 30 days in advance of submission in order to obtain approval.